CLINICAL TRIAL: NCT00003086
Title: Phase I/II Study of Samarium 153 as Part of a Double (Sequential) Autologous Bone Marrow Transplant (ABMT) for Patients With Stage IV Breast Cancer
Brief Title: Repeated Bone Marrow Transplantation in Treating Women With Advanced Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: no participants enrolled in a three year period
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: LSU-97447; CDR0000065786 (Registry Identifier: PDQ (Physician Data Query)); NCI-V97-1341
Record Dates: First submitted 1999-11-01; First posted 2004-02-09 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; CAF protocol; Carboplatin; Cisplatin; Cyclophosphamide; Doxorubicin; Fluorouracil; Ifosfamide; Melphalan; Paclitaxel; Thiotepa; Peripheral Blood Stem Cell Transplantation; samarium Sm-153 lexidronam

INTERVENTIONS:
Biological: filgrastim
Drug: CAF regimen
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: fluorouracil
Drug: ifosfamide
Drug: melphalan
Drug: paclitaxel
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation
Radiation: samarium Sm 153 lexidronam pentasodium

SUMMARY:
RATIONALE: Bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of repeated use of high-dose chemotherapy plus bone marrow transplantation and samarium 153 in treating women who have stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) of samarium 153 used sequentially with autologous bone marrow transplantation for metastatic breast cancer. II. Determine the response rate, median duration of response, and overall survival of patients who respond to induction therapy followed by 2 cycles of high dose chemotherapy and stem cell support.

OUTLINE: This is a dose escalation study. Patients are first treated with salvage chemotherapy for no more than 4 cycles. At least a partial remission must be achieved. Peripheral blood stem cells (PBSC) are collected following the administration of filgrastim (granulocyte colony-stimulating factor; G-CSF). After recovery from the prior chemotherapy, high dose chemotherapy begins. Paclitaxel is administered as a 24 hour infusion on day -7. Melphalan IV is administered over 1 hour on days -6 and -5. PBSC are infused on day 0. A second regimen of high dose chemotherapy begins after at least 42 days posttransplant and as long as at least partial remission occurs after previous chemotherapy. Samarium 153 is administered on day -14. Cohorts of 3 patients each are treated at each dose level until the maximum tolerated dose is reached (defined as dose at which the dose limiting toxicity occurs in 3 or more of 6 patients). Cyclophosphamide, thiotepa, and carboplatin are infused over 24 hours on days -7 through -4. PBSC are infused on day 0 followed by G-CSF IV. The phase II dose of samarium 153 is one dose level below the MTD determined in the Phase I portion of this study. Patients are followed until death.

PROJECTED ACCRUAL: At least 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic breast cancer Adequate peripheral blood stem cells harvested and stored

PATIENT CHARACTERISTICS: Age: 21-65 Sex: Female Performance status: 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 1.5 mg/dL SGOT and SGPT normal Renal: Creatinine less than 1.5 mg/dL Cardiovascular: Ejection fraction of at least 50% No symptomatic coronary artery disease Pulmonary: FEV1 and DLCO greater than 50% of predicted Other: Not pregnant Not HIV positive Not hepatitis B surface antigen positive No uncontrolled infection No other prior malignancy within 5 years except: Curatively treated in situ adenocarcinoma of the cervix Curatively treated nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY: Recovered from toxic effects of prior therapy Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for metastatic disease Prior adjuvant chemotherapy allowed Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for metastatic disease Surgery: Not specified

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 1997-03; Primary Completion 2001-01-28 (Actual); Study Completion 2001-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin B. Weinberger, MD, Study Chair — Feist-Weiller Cancer Center at Louisiana State University Health Sciences
Locations (1):
- Louisiana State University School of Medicine, Shreveport, Louisiana, United States